CLINICAL TRIAL: NCT04991246
Title: Project FLUx COntact-CoVID-19 Faculty of Medicine Paris-Saclay
Acronym: FLUCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP210403; 2021-A00663-38 (Other: IDRCB)
Record Dates: First submitted 2021-07-05; First posted 2021-08-05 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: Simulation; epidemiology; public health; computer science; infectiology; technology; pandemic COVID
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Students, teachers,administrative staff from the medical school of Paris-Saclay University (Experimental): Students,teachers,administrative staff from the medical school of Paris-Saclay University
  Interventions: Other: Antigenic tests (on saliva samples); Other: Individual electronic sensor port; Other: Atmospheric measurements of CO2

INTERVENTIONS:
Other: Antigenic tests (on saliva samples) — SARS-CoV-2 screening tests: two massive antigenic tests campaigns (on salivary samples).
Other: Individual electronic sensor port — Individual electronic sensor recording contacts but not their location (in the form of a bracelet, a key ring or a badge) Contact data collection points (5 maximum, located at compulsory passage points for participants). When a sensor is close to one of these terminals, it discharges its contacts in seconds.
Other: Atmospheric measurements of CO2 — Atmospheric measurements of CO2 in the relevant closed places of the faculty (lectures / practical work / BU / refectory): battery operated sensors. When a sensor is installed in a place, the ventilation conditions (number of open windows, etc.) as well as the number of people present will be noted.

SUMMARY:
The worldwide health system has been marked by the SARS-CoV-2 pandemic. French educational system has been upset, especially medical schools, which, because of their hospital location, are particularly exposed to the spread of the virus. The medical school of Paris-Saclay University, located within bicetre University Hospital, AP-HP, must therefore adapt on a daily basis to ensure educational continuity. Taking advantage of an exceptional scientific ecosystem, innovative viral epidemic propagation modeling approaches based on both simulation and contact tracing data will be tested in real-life conditions. These propagation models will serve to scientifically optimize future educational organization procedures in this medical school.

DETAILED DESCRIPTION:
All the participants will be equipped with individual wireless contact tracing technology. Anonymised contact events will be automatically monitored for a period of two months to measure the daily contact flow density between the students at medical school. Epidemic simulation models will be enriched with these real contact tracing data to generate optimized viral propagation probability networks. During the same period, CO2 measurement will be performed in several relevant sectors (classrooms, amphitheaters, corridors etc) to allow a more holistic understanding of the propagation conditions. Finally, the probabilistic models will be confronted to the results of a two step COVID-19 screening campaign.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of adult men and women over 18 from the Paris-Saclay Medicine UFR

  * Belonging to the teaching staff
  * Belonging to the promotions of DFGSM 2 and 3, and DFASM 1 and 2 (2nd to 5th year of medical study)
  * administrative staff
* Affiliated to a social security scheme or beneficiary (excluding AME)
* Informed and written consent

Exclusion Criteria:

* Absence of intercurrent disease before inclusion
* Positive antigenic or PCR test at the time of inclusion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Simulations results compared with the COVID-19 two-step screening campaign results | 2 months
  Develop and validate a simulation tool for the spread of an epidemic in a university-type environment, updated by the effective measurement of contacts between individuals (wireless digital search of contacts).

SECONDARY OUTCOMES:
CO2 atmospheric measurement | 2 months
  The CO2 rate will be measured under very diverse conditions in terms of room size, number of people, type of ventilation. These systematic measurements together with the reading of precise conditions will allow us to establish a precise correspondence between the various factors and this rate. This should improve our understanding of the chains of contamination. and the circumstances that may have favored the spread of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier LAMBOTTE, Pr, Principal Investigator — Bicetre Hospital
Locations (1):
- CHU Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No